CLINICAL TRIAL: NCT00353119
Title: Phase 3 Study With a Placebo-Controlled, Double-blind, on the Safety and Efficacy of Etanercept in Palmo-Plantar Pustulosis
Brief Title: A Placebo-Controlled Double-Blind Study on the Safety and Efficacy of Etanercept in Palmoplantar Pustulosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2.3
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Results first posted 2010-12-21 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Palmoplantaris Pustulosis
Keywords: Palmoplantar pustulosis; Psoriasis; Etanercept
MeSH Terms: conditions — Psoriasis | interventions — Sodium Chloride; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo then etanercept (Placebo Comparator): Patients randomized to initiate the study with placebo for the first 12 weeks - Group 1 then crossed over to etanercept 50mg twice weekly for weeks 12 to 24
  Interventions: Drug: Placebo comparator; Drug: Etanercept
- Etanercept (Active Comparator): Patients randomized to etanercept - Group 2. Patients received etanercept 50 mg subcutaneously twice weekly for 24 weeks
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Placebo comparator — Patients received placebo subcutaneously twice weekly
  Other Names: Saline
  Arms: Placebo then etanercept
Drug: Etanercept — Patients received etanercept 50 mg subcutaneously twice weekly
  Other Names: Enbrel

SUMMARY:
Palmoplantar pustulosis (PPP) is a chronic recurrent skin condition characterized by the presence of pustules, erythema and hyperkeratosis on palms and soles. PPP can be a severe and disabling disease limiting the ability to walk or work. Although studies on the quality of life of patients with PPP are not available, a recent investigation showed that palmoplantar psoriasis (non pustular) has a more important impact on quality of life than plaque psoriasis. This important impact on quality of life is not surprising as palmoplantar psoriasis as well as palmoplantar pustulosis may limit the ability to work or conduct activities with hands or even impair walking. The disease is sometimes associated with psoriasis elsewhere on the body. Current treatments for PPP include topical corticosteroids, cyclosporine, PUVA therapy, methotrexate and acitretin. Response to topical corticosteroids and PUVA therapy is often disappointing presumably because the thickness of the stratum corneum on palms and soles prevents good penetration of topical medications and light. Cyclosporine and methotrexate are sometimes used with success for PPP but there are concerns with long term toxicity of both drugs. Therefore there is a need for new treatments for PPP.

DETAILED DESCRIPTION:
This is a placebo-controlled double blind study. Patients will be randomized to receive etanercept versus placebo in a 2:1 fashion for the first 3 months. All patients will receive etanercept in the last 3 months.

Patients with active PPP will be included. A washout of 4 weeks for systemic medications and 2 weeks for Psoralen Ultra Violet A (PUVA) therapy will be required. A washout period of 2 weeks will be required for all other topical medications. The Palmoplantar pustulosis severity index (PPPASI) will be used to evaluate severity. Only patients with a severity score of 8 or more on hands and/or feet will be included. Safety will be assessed by performing physical examinations, evaluation of adverse events and biological parameters (complete blood count (CBC), chemistry, urinalysis).

High quality digital medical photographs will be taken at baseline, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Palmoplantar pustulosis with a severity score of at least 8 on hands and-or feet
* Age 18 years or older
* Patient who would benefit from systemic therapy
* Unless surgically sterile (or at least 1 year post-menopausal for women) patients (heterosexual men and women) must have used a effective method of contraception for at least 30 days before the start of the study drug and until at least 1 month after the last drug administration
* Informed consent obtained
* Normal or non clinically significant chest X ray taken within 6 months of screening
* Negative serum pregnancy test at screening and negative urine pregnancy test at day 0 for women of childbearing potential
* Negative personal history of tuberculosis
* Presence of PPP for more than 6 months
* Subject must be willing to inject themselves subcutaneously.
* Negative PPD results

Exclusion Criteria:

* Use of topical steroids, topical tar preparations, or other topical anti PPP or anti-psoriatic preparations within the past two weeks
* Unstable forms of psoriasis (acute guttate psoriasis, psoriatic erythroderma, generalized pustular psoriasis)
* At the investigator's discretion any significant infection within 30 days of screening or a patient at risk of septicemia
* Presence of acute forms of tinea pedis and other causes of pustular eruptions of the palms and soles apart from PPP based on clinical evaluation
* Evidence of any skin condition that would interfere with the evaluation of PPP
* Use of investigational drugs within the past four weeks
* Use of systemic anti-PPP or anti-psoriatic drugs such as steroids, retinoids, or methotrexate within the past four weeks
* Use of parenteral systemic antibiotics within the past four weeks
* Use of cyclosporine within the past four weeks
* Use of ultraviolet light therapy (UVB, nbUVB or PUVA) within the past two weeks
* An unstable or serious medical condition
* Known sero-positivity for the HIV virus
* Known hypersensitivity to etanercept or one of its components
* Receipt of live attenuated vaccines 12 weeks or less before Day 0 and during the course of the study
* Pregnant or breast feeding female subject
* Any significant medical condition that might cause this study to be detrimental to the patient
* At the investigator's discretion current or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
* Presence of congestive heart failure
* Presence of a demyelinating disorder (optic neuritis, multiple sclerosis or other)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD MSc FRCPC, Principal Investigator — Innovaderm Research Incorporated
Locations (3):
- Canada (3):
  - Innovaderm Research Incorporated, Laval, Quebec
  - Innovaderm Research Incorporated, Montreal, Quebec
  - Centre de Recherche Dermatologique du Québec métropolitain, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Period: First Intervention Day 0 to Week 12
Arm/Group | Placebo Then Etanercept | Etanercept
Started | 5 | 10
Completed | 5 | 10
Not Completed | 0 | 0
Period: Second Intervention Week 12 to Week 28
Arm/Group | Placebo Then Etanercept | Etanercept
Started | 5 | 10
Completed | 5 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Etanercept | Etanercept | Total
Number analyzed (Participants) | 5 | 10 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 15
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 54.2 (4.76) | 46.9 (13.3) | 49.33 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 10 | 15
PPPASI - Palmoplantar Pustulosis Area and Severity Index [Mean (Standard Deviation); unit: Units on a scale] — PPPASI = (E + I + D)Area X 0.2 (R palm) + (E + I + D) Area X 0.2 (L palm) + (E + I + D) Area X 0.3 (R sole) + (E + I + D) Area X 0.3 (L sole).
  Erythema, induration and desquamation are evaluated on a scale of 0 to 4 while area is evaluated on a scale of 0 to 6. The m-PPPASI score can vary from 0 (absence of disease) to 72 (most severe palmoplantar psoriasis possible).
  Units on a scale | 21.3 (10.3) | 16.3 (5.0) | 18.0 (7.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Palmoplantar Pustulosis Severity Index (PPPASI) Before Crossover
Description: Comparison of the percentage change in Palmoplantar pustulosis severity index PPPASI) at 12 weeks in patients treated with placebo or etanercept
  PPPASI = (E + I + D)Area X 0.2 (R palm) + (E + I + D) Area X 0.2 (L palm) + (E + I + D) Area X 0.3 (R sole) + (E + I + D) Area X 0.3 (L sole).
  Erythema, pustules and desquamation are evaluated on a scale of 0 to 4 while area is evaluated on a scale of 0 to 6. The PPPASI score can vary from 0 (absence of disease) to 72 (most severe palmoplantar psoriasis possible).
Time Frame: 12 weeks
Population: The intent to treat (ITT) population is the same as the per protocol (PP) population. There was no imputation technique necessary.
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- Placebo: Patients randomized to initiate the study with placebo for the first 12 weeks - Group 1
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 5 | 10
Percentage change | 30.1 (25.7) | 7.1 (60.4)

2. Secondary Outcome: Number of Adverse Events
Description: Study the safety of etanercept in patients with PPP by collecting adverse events from the screening visit until week 28. For a given AE, a subject will be counted once even if he or she has experienced multiple episodes for that particular AE. An adverse event is any untoward medical occurrence including any clinically significant abnormal laboratory values or variation from the baseline condition to the last visit (week 28) in a patient receiving a pharmaceutical product, without regards to the possibility of a causal relationship with this treatment.
Time Frame: 28 weeks
Population: Patients that crossed over from placebo to etanercept are included in the Etanercept group. The placebo group only included adverse events from the first 12 weeks prior to the crossover. The intent to treat (ITT) population is the same as the per protocol (PP) population. There was no imputation technique necessary.
Measure: Number; unit: Adverse Events
Groups:
- Etanercept: Patients randomized to etanercept - Group 2. Patients received etanercept 50 mg subcutaneously twice weekly for 24 weeks AND Patients that crossed over to etanercept 50 mg subcutanously twice weekly after taking placebo for the first 12 weeks.
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 5 | 15
Adverse Events | 13 | 57

3. Secondary Outcome: Percentage Change in Palmoplantar Pustulosis Area and Severity Index (PPPASI)
Description: Evaluate efficacy using palmoplantar pustulosis area and severity index (PPPASI) in patient with palmoplantar pustulosis treated with etanercept for 6 months
  PPPASI = (E + I + D)Area X 0.2 (R palm) + (E + I + D) Area X 0.2 (L palm) + (E + I + D) Area X 0.3 (R sole) + (E + I + D) Area X 0.3 (L sole).
  Erythema, pustules and desquamation are evaluated on a scale of 0 to 4 while area is evaluated on a scale of 0 to 6. The PPPASI score can vary from 0 (absence of disease) to 72 (most severe palmoplantar psoriasis possible).
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Etanercept
Number analyzed (Participants) | 10
Percentage change | 30.1 (36.1)

4. Secondary Outcome: Percentage Change in Palmoplantar Pustulosis Area and Severity Index (PPPASI) After Crossover
Description: as for outcome 3
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- Etanercept After Placebo: Group 1 patients that crossed over to etanercept 50mg twice weekly for weeks 12 to 24 after having initiated the study with placebo for the first 12 weeks
Arm/Group | Etanercept After Placebo
Number analyzed (Participants) | 5
Percentage change | 52.1 (15.4)

ADVERSE EVENTS:
Groups:
- Placebo: Patients randomized to initiate the study with placebo for the first 12 weeks
- Etanercept: Patients randomized to etanercept who received etanercept 50 mg subcutaneously twice weekly for 24 weeks AND patients who crossed over to etanercept 50 mg subcutaneously twice a week for 12 weeks.
Arm/Group | Placebo | Etanercept
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/10
Other Adverse Events (participants affected / at risk) | 5/5 | 15/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | Etanercept (N=15)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bilateral burning both feet (Nervous system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Candida Vaginitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Common Cold (Infections and infestations) | 2 (2) | 4 (6)
Dental Extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Diahhrea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Erythema to thighs (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flu (Infections and infestations) | 0 (0) | 1 (1)
General Malaise (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 4 (4)
Hematoma (Vascular disorders) | 0 (0) | 1 (2)
Herpes Labialis (Infections and infestations) | 1 (1) | 1 (2)
Increase in arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Increase in depression (Psychiatric disorders) | 0 (0) | 1 (1)
Increase in psoriatic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 10 (14)
Intermitant uticaria crisis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mild leucocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Occasional spotting (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Occult hematuria (Investigations) | 0 (0) | 1 (1)
Pain thoracic wall (General disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Positional vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pruritus under both feet (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tendinitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (2) | 0 (0)
Wisdom tooth pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Worsening of feet plantar pustulosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: embargo of 60 days or less